CLINICAL TRIAL: NCT02080845
Title: Effects of a Cocoa Shot on the Human Brain 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: The Hershey Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB00026868
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Caffeine
Keywords: Caffeine; MRI; Brain blood flow; Cognition; Perfusion; Resting functional magnetic resonance imaging (fMRI)
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- no caffeine & no theobromine (Placebo Comparator): Drink 1
  Interventions: Dietary Supplement: no caffeine; Dietary Supplement: no theobromine
- no caffeine & low theobromine (Experimental): Drink 2
  Interventions: Dietary Supplement: no caffeine; Dietary Supplement: low theobromine
- no caffeine & high theobromine (Experimental): Drink 3
  Interventions: Dietary Supplement: no caffeine; Dietary Supplement: high theobromine
- high caffeine & no theobromine (Experimental): Drink 4
  Interventions: Dietary Supplement: high caffeine; Dietary Supplement: no theobromine

INTERVENTIONS:
Dietary Supplement: no caffeine
  Arms: no caffeine & high theobromine; no caffeine & low theobromine; no caffeine & no theobromine
Dietary Supplement: high caffeine
  Arms: high caffeine & no theobromine
Dietary Supplement: no theobromine
  Arms: high caffeine & no theobromine; no caffeine & no theobromine
Dietary Supplement: low theobromine
  Arms: no caffeine & low theobromine
Dietary Supplement: high theobromine
  Arms: no caffeine & high theobromine

SUMMARY:
The Hershey Company is interested in investigating the effects of various chocolate beverages on brain physiology and cognitive function. The main substances in the drinks that are known to influence the brain are caffeine and related chemicals such as theobromine. Caffeine and chemicals related to caffeine are all naturally occurring and all potentially alter brain physiology. This study will evaluate changes in brain blood flow and cognition following the consumption of drinks with various combinations of the Primary Ingredients. The study proposed here will evaluate ingredients in a 4-arm cross-over double-blind design in an attempt to understand the differential effects of these compounds in chocolate drinks.

ELIGIBILITY:
Inclusion Criteria:

* Consume 200-500 mg caffeine daily
* Willing and capable of signing the informed consent
* Willing to attend 4 testing sessions that will take 4-6 hours each AND will be at least 10 days apart
* Willing to abstain from caffeine for 16 hours before each testing session
* Willing to and able to have MRIs

Exclusion Criteria:

* As determined from the medical screening session

  * active neurological dysfunction (such as a major Axis I psychopathology, Alzheimer's disease, Parkinson's disease, prior history of stroke, epilepsy, or serious central nervous system (CNS) trauma)
  * attention deficit hyperactivity disorder (ADHD)
  * migraines
  * hypertension
  * diabetes
  * peripheral vascular disease
  * taking vasoactive medications (such as anti-hypertensive medications)
  * depression that has not been on a stable medical treatment for at least 4 weeks
  * Pregnancy
  * Allergy to chocolate, peanuts, tree nuts, egg, soy, milk, wheat
* Color blindness
* Individuals who are or potentially may be cognitively or psychologically impaired, or who otherwise have a limited capacity to provide consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-03; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in Working Memory (% correct) | Baseline, 1.5 hour and 3.5 hours post beverage
  N-Back Task
Change in Response Time (milliseconds) | Baseline, 1.5 hour and 3.5 hours post beverage
  Choice ResponseTime Task
Change in Short Term Memory (# correct) | Baseline, 1.5 hour and 3.5 hours post beverage
  Hopkins Verbal Learning Task (HVLT)
Change in Mood (change in Likert scale score) | Baseline, 1.5 hour and 3.5 hours post beverage
  Profile of Mood Status (POMS)
Change in Attention (% accuracy) | Baseline, 1.5 hour and 3.5 hours post beverage
  Eriksen Flanker Task
Change in Executive Function (# correct) | Baseline, 1.5 hour and 3.5 hours post beverage
  Stroop Task

SECONDARY OUTCOMES:
Change in Brain Blood Flow (ml/g/min) | 1 hour post beverage
  Non-invasive brain perfusion measured with arterial spin labeling magnetic resonance imaging
% Change in Heart Rate (beats/minute) | before, 1 hour, and 3 hour post beverage
  Pulse
% Change in Blood Pressure (mm Hg) | before, 1 hour, and 3 hour post beverage
Change in Respiration (breaths/minute) | before, 1 hour, and 3 hour post beverage

OTHER OUTCOMES:
% Change in Brain Connectivity (network degree) | 1 hour post beverage
  Measures of functional brain connectivity based on resting-state functional magnetic resonance imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Laurient, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States